CLINICAL TRIAL: NCT01814696
Title: The Effect of the MedSentry System on Medication Adherence for Patients With Congestive Heart Failure: A Pilot Study
Brief Title: The Effect of the MedSentry System on Medication Adherence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment and reached number needed for analysis.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-P-002181
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Congestive Heart Failure; Medication Adherence; Medication Compliance; Telemedicine; Telehealth
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Subjects will continue to receive usual medical care from their doctor(s).
- MedSentry System (Experimental): Subjects will continue to receive usual medical care from their doctor(s). Subjects will use the MedSentry System and electronic pillbox, to manage their medications.
  Interventions: Device: MedSentry System

INTERVENTIONS:
Device: MedSentry System — Subjects will use the MedSentry System and electronic pillbox, to manage their medications.
  Other Names: MedSentry pillbox; Electronic pillbox; Pillbox
  Arms: MedSentry System

SUMMARY:
The goal of this pilot study to evaluate the effect of the MedSentry system, a multi-faceted medication adherence device and reminder system, on medication adherence and clinical outcomes in heart-failure (HF) patients. We will also evaluate the usability and satisfaction derived from using this system.

We hypothesize that:

1. The use of the MedSentry system will improve medication adherence in patients with a discharge diagnosis of HF.
2. The improvement in adherence correlates with fewer hospitalizations and emergency department (ED) visits.
3. The improvement in adherence correlates with better health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed the Partners Connected Cardiac Care Program (CCCP)
* Take at least 3 and no more than 10 different daily medications (including both prescription and non-prescription/over the counter medications) to treat Heart Failure (HF) and other comorbid disorders.
* Take medications no more than 4 specified times each day (i.e. morning, afternoon, early evening, bedtime).
* The patient must be able to open a pill bottle independently.
* The patient must be able to sort and manage their own medications.
* Hospitalization within the last 24 months.
* Have a telephone or cell phone.
* Live in the greater Boston area.
* The patients must speak, read and write English.
* The patients must not be either vision or hearing impaired (i.e., unable to hear an alarm similar to a clock alarm or oven alarm).
* Patient must have an Massachusetts General Hospital (MGH) affiliated care provider.

Exclusion Criteria:

* Dementia or other conditions precluding the participant from providing informed consent or from learning to use the MedSentry pillbox.
* Home environment unsuitable for the MedSentry pillbox and other installed equipment.
* Awaiting revascularization, cardiac resynchronization or heart transplant.
* Patients with a coexisting terminal illness like cancer or Chronic Renal Failure (CRF) requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hale TM, Jethwani K, Kandola MS, Saldana F, Kvedar JC. A Remote Medication Monitoring System for Chronic Heart Failure Patients to Reduce Readmissions: A Two-Arm Randomized Pilot Study. J Med Internet Res. 2016 Apr 17;18(5):e91. doi: 10.2196/jmir.5256. PMID 27154462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a list of HF patients who had successfully completed a HF telemonitoring program at Massachusetts General Hospital (MGH) or Brigham & Women's Hospital (BWH) and had been hospitalized in the previous 24 months.
Groups:
- Control: Subjects will continue to receive usual medical care from their doctor(s).
  Subjects will follow their normal medication management routine.
- Intervention: Subjects will continue to receive usual medical care from their doctor(s).
  Intervention: Subjects will use the MedSentry System and electronic pillbox, to manage their medications.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 15 | 11
Completed | 13 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Randomized to wrong group | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Subjects will continue to receive usual medical care from their doctor(s). Subjects will use the MedSentry System and electronic pillbox, to manage their medications.
  MedSentry System: Subjects will use the MedSentry System and electronic pillbox, to manage their medications.
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (10.4) | 68.4 (11.8) | 71.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 9 | 7 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 9 | 22
  Non-White | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25
Marital Status [Number; unit: participants]
  Married | 7 | 4 | 11
  Non-married | 7 | 7 | 14
Lives Alone [Number; unit: participants]
  Lives Alone | 6 | 4 | 10
  Lives with Others in Household | 8 | 7 | 15
Education Level [Number; unit: participants]
  Less than 1 year college | 3 | 4 | 7
  1 or more years of college | 11 | 7 | 18
Internet User [Number; unit: participants]
  Internet User | 10 | 6 | 16
  Non-Internet User | 4 | 5 | 9
Mobile Phone Ownership [Number; unit: participants]
  No mobile phone | 1 | 2 | 3
  Cellphone | 11 | 7 | 18
  Smartphone | 2 | 2 | 4
Medical Outcomes Study (MOS) Adhere [Number; unit: participants] — Single Medication Adherence Measures, Medical Outcomes Study (MOS) "Adhere"
  participants
    Adherent | 11 | 7 | 18
    Non-adherent | 3 | 4 | 7
Using a Medication Reminder Tool [Number; unit: participants]
  Using a medication reminder | 11 | 7 | 18
  Not using a medication reminder | 3 | 4 | 7
NYHA Functional Classification [Number; unit: participants] — This scale is a categorical measure of severity of heart failure. There are four categories ranging from 1-4 increasing in severity.
  participants
    Class 1 | 11 | 1 | 12
    Class 2 | 1 | 9 | 10
    Class 3 | 1 | 1 | 2
    Class 4 | 0 | 0 | 0
    Unknown | 1 | 0 | 1
Self-Rated Health [Number; unit: participants]
  Poor | 0 | 1 | 1
  Fair | 6 | 5 | 11
  Good | 5 | 5 | 10
  Very Good | 2 | 0 | 2
  Excellent | 1 | 0 | 1
Personal Health Questionnaire Depression Scale, 8-Items (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — The PHQ-8 is a commonly used measure of depression. Each of the 8-items is scored from 0 to 3 to generate a total score from 0 to 24. Generally accepted cut points for depression severity are 5-9 = mild, 10-14 = moderate, 15-19 = moderately severe, and 20-24 = severe.
  units on a scale | 3.5 (4.6) | 6.8 (4.5) | 5.0 (4.8)
Minnesota Living with Heart Failure Questionnaire (MLHFQ) Total Score [Mean (Standard Deviation); unit: units on a scale] — Health-related quality of life is measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The questionnaire consists of 21 items that assess the impact of HF and HF treatment on key physical, emotional, and social dimensions of a patient's life during the past four weeks. Responses are coded from 0 = does not apply and 1 = very little to 5 = very much.
  A higher score represents a greater negative HR-related impact on quality of life.
  units on a scale | 26.2 (23.1) | 43.7 (25.9) | 34.3 (25.6)
Minnesota Living with Heart Failure Questionnaire (MLHFQ) Physical Score [Mean (Standard Deviation); unit: units on a scale] — Health-related quality of life is measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The Physical Sub-scale is created from 8-items from the 21-items that make up the MLHFQ. The items assess the impact of HF and HF treatment on key physical dimensions of a patient's life during the past four weeks. Responses are coded from 0 = does not apply and 1 = very little to 5 = very much.
  The sub-scale ranges in possible values from 0 to 40. A higher score represents a greater negative HR-related impact on quality of life.
  units on a scale | 10.8 (11.4) | 21.9 (11.8) | 15.7 (12.7)
Minnesota Living with Heart Failure Questionnaire (MLHFQ) Emotional Score [Mean (Standard Deviation); unit: units on a scale] — Health-related quality of life is measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The Emotional Sub-scale is created from 5-items from the 21-items that make up the MLHFQ. The items assess the impact of HF and HF treatment on key emotional dimensions of a patient's life during the past four weeks. Responses are coded from 0 = does not apply and 1 = very little to 5 = very much.
  The sub-scale ranges in possible values from 0 to 25. A higher score represents a greater negative HR-related impact on quality of life.
  units on a scale | 5.9 (6.2) | 7.2 (7.7) | 6.5 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Medical Outcomes Study (MOS) "Adhere"
Description: Subject reported medication adherence. The Medical Outcomes Study (MOS) "Adhere" medication adherence measure consists of a single question that asks participants "How often did you take your medications as prescribed during the past 4 weeks?" Responses are recoded into a dichotomous measure of nonadherent (none, a little, some of the time) and adherent (most, all of the time).
Time Frame: 3 months
Population: Participants who completed questions on enrollment and closeout survey.
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 13 | 11
participants
  Adherent | 9 | 8
  Non-adherent | 4 | 3
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.605, Fisher Exact — a prior threshold p<0.05

2. Secondary Outcome: Number of Participants With 1 or More Emergency Department (ED) Visits.
Time Frame: 3 months
Population: Intention to treat analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 14 | 11
participants
  Heart Failure Related | 3 | 1
  Non Heart Failure Related | 4 | 3
  All Cause | 7 | 4
Statistical Analysis 1: Comparison: Control vs Intervention; Heart failure related ED visits; Test type: Superiority or Other; p = 0.604, Fisher Exact
Statistical Analysis 2: Comparison: Control; Non-heart failure related ED visits; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Control vs Intervention; All cause ED visits; Test type: Superiority or Other; p = 0.677, Fisher Exact

3. Secondary Outcome: Number of Participants With 1 or More Hospitalizations.
Time Frame: 3 months
Population: Intention to treat analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 14 | 11
participants
  Heart Failure Related | 4 | 1
  Non Heart Failure Related | 4 | 1
  All Cause | 7 | 1
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.341, Fisher Exact
Statistical Analysis 2: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.042, Fisher Exact

4. Secondary Outcome: Number of Emergency Department (ED) Visits.
Time Frame: 3 months
Population: Intention to treat analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 14 | 11
participants
  All cause | 7 | 4
  Heart Failure Related | 3 | 1
  Non Heart Failure Related | 4 | 3
Statistical Analysis 1: Comparison: Control vs Intervention; All cause; Test type: Superiority or Other; p = 0.497, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Control vs Intervention; Heart failure related; Test type: Superiority or Other; p = 0.413, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Control vs Intervention; Non-heart failure ED visits; Test type: Superiority or Other; p = 0.944, Wilcoxon rank-sum test

5. Secondary Outcome: Number of Hospitalization Visits.
Time Frame: 3 months
Population: Intention to treat analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 14 | 11
participants
  All cause | 8 | 2
  Heart Failure Related | 4 | 1
  Non Heart Failure Related | 4 | 1
Statistical Analysis 1: Comparison: Control vs Intervention; All cause; Test type: Superiority or Other; p = 0.057, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Control vs Intervention; Heart failure related; Test type: Superiority or Other; p = 0.236, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Control vs Intervention; Non heart failure related; Test type: Superiority or Other; p = 0.236, Wilcoxon rank-sum test

6. Secondary Outcome: Hospitalization, Length of Stay (Days)
Time Frame: 3 months
Population: Intention to treat analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 14 | 11
days
  All cause | 2.34 (3.13) | 0.36 (1.21)
  Heart Failure Related | 1.36 (2.68) | 0.18 (0.60)
  Non Heart Failure Related | 1.07 (2.06) | 0.18 (0.60)
Statistical Analysis 1: Comparison: Control vs Intervention; All cause; Test type: Superiority or Other; p = 0.034, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Control vs Intervention; Heart failure related; Test type: Superiority or Other; p = 0.196, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Control vs Intervention; Non heart failure related; Test type: Superiority or Other; p = 0.210, Wilcoxon rank-sum test

7. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire (MLHFQ) Total Summary Score
Description: Health-related quality of life is measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). The questionnaire consists of 21 items that assess the impact of HF and HF treatment on key physical, emotional, and social dimensions of a patient's life during the past four weeks. Responses are coded from 0 = does not apply and 1 = very little to 5 = very much.
  A higher score represents a greater negative HR-related impact on quality of life.
Time Frame: Baseline, end 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 13 | 11
units on a scale | 28.2 (22.3) | 62.2 (20.6)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse Events were categorized as cardiac and non-cardiac types.
  Adverse Events classified as cardiac types during the study included: angina; wide complex tachycardia; automatic implantable automatic defibrillator firing; endocarditis; and dizzy, low blood pressure. Adverse Events classified as non-cardiac types during this study included: fell; cellulitis; confusion; fever, shortness of breath, asthma; and ear pain.
Arm/Group | Control | Intervention
Serious Adverse Events (participants affected / at risk) | 7/14 | 3/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=14) | Intervention (N=11)
ED Visit (Cardiac disorders) | 3 (3) | 1 (1)
ED Visit (General disorders) | 4 (4) | 3 (3)
Hospitalization (Cardiac disorders) | 4 (4) | 1 (1)
Hospitalization (General disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
The initial goal was to enroll a total of 70 participants with 35 randomized to each of the two study arms. However, due to slow enrollment the study was ended early with 26 participants having completed enrollment and randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No